CLINICAL TRIAL: NCT07201194
Title: HOL-AKU: Holistic Acupuncture for Patients With Chemotherapy Induced Nausea
Brief Title: Holistic Acupuncture for Patients With Chemotherapy Induced Nausea
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vejle Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: HOL-AKU
Record Dates: First submitted 2025-09-23; First posted 2025-10-01 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer; Prostate Cancer; Lung Cancer; Gynaecologic Cancer; Colorectal Cancer; Pancreatic Cancer Metastatic
Keywords: acupuncture; chemotherapy induced nauseau
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms; Lung Neoplasms; Colorectal Neoplasms | interventions — Acupressure

STUDY DESIGN:
Intervention Model Description: The project employs a crossover design, in which the patients participate in both the intervention and the control group. Participants are randomized into two groups: one group receives the intervention first and subsequently serves as the control group, while the other group starts as the control and later receives the intervention.
  Based on a holistic and individualized consultation, participants in the intervention group will receive one treatment with holistic acupuncture and acupressure in connection with a standard chemotherapy session, including standard supportive care for nausea. The control group will receive standard chemotherapy and supportive care only.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Holistic acupuncture and acupressure (Experimental): Holistic acupuncture and acupressure as a supplement to standard care
  Interventions: Other: Holistic acupuncture and acupressure
- Standard care (Active Comparator)
  Interventions: Other: Standard medical treatment

INTERVENTIONS:
Other: Holistic acupuncture and acupressure — The intervention consists of one holistic and individualized consultation with an oncologist trained in acupuncture, in connection with outpatient chemotherapy. The consultation follows the principles of Traditional Chinese Medicine (TCM). The theoretical framework applied is Zang-Fu, which describes organ imbalances and aligns closely with Western medical understanding.
  Based on individual assessment and anamnesis, the patient receives acupuncture combined with acupressure.
  A maximum of 10 needles will be used, regardless of whether a deficiency or excess condition is identified. The acupuncture needles used are CAIR Super Silicon CSC-1, size 0.20 × 25 mm. The needles are inserted perpendicularly, except for Yin Tang, which is inserted transversely. The needles will remain in place for 25 minutes.
  Arms: Holistic acupuncture and acupressure
Other: Standard medical treatment — Standard treatment and care includes chemotherapy, supportive antiemetic medication, close monitoring, and management of the patient's symptoms, side effects, and overall health.
  Arms: Standard care

SUMMARY:
The study explores whether acupuncture as a supplement to conventional antiemetic medicine is superior in reducing the level of chemotherapy induced nausea compared to conventional anitemetic medicine alone.

A total of 90 patients experiencing chemotherapy induced nausea will be allocated 1:1 to either acupuncture and antiemetic medicine or antiemetic medicine alone.

The level of nausea and other cancer related symptoms will be assessed at baseline and 8 and 22 days after enrollment

ELIGIBILITY:
Inclusion criteria

* ≥ 18 years of age
* Undergoing chemotherapy and experiencing nausea despite adherence to the prescribed antiemetic regimen
* Understands and speaks Danish
* Written and orally informed consent
* Planned for treatment every 14 days
* At least two chemotherapy cycles planned at the time of inclusion

Exclusion Criteria:

* Brain metastases
* Performance status >2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-11-17 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient reported nausea assessed on the EORTC-15-PAL Scale | 8 days after enrollment

SECONDARY OUTCOMES:
Patient reported symptom intensity according to the EORTC-15 PAL Scale | 8 and 22 days after enrollment

OTHER OUTCOMES:
Patient reported use of antiemetic medicine | 8 and 22 days after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Mette Stie, Phd, Principal Investigator — Department of Oncology, Lillebaelt Hospital, Vejle
Locations (1):
- Department of Oncology, Vejle Hospital, Vejle, Denmark

IPD SHARING:
Plan to Share IPD: No